CLINICAL TRIAL: NCT04066998
Title: Cytokine Profile of Conjunctivitis, Performed Through Tears Analysis Among Patients Treated With Dupilumab
Acronym: CYCLADDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P/2019/424
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-08

CONDITIONS: Conjunctival Diseases; Atopic Dermatitis; Side Effect
MeSH Terms: conditions — Conjunctival Diseases; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conjunctivitis (Experimental): Patients treated with Dupilumab with conjunctivitis
  Interventions: Other: Tears sampling; Other: Lashes sampling
- No conjunctivitis (Other): Patients treated with Dupilumab and showing no signs of ocular involvement
  Interventions: Other: Tears sampling; Other: Lashes sampling

INTERVENTIONS:
Other: Tears sampling — Tears sampling
Other: Lashes sampling — Lashes sampling

SUMMARY:
This study aims to assess the cytokine profile of tears in patients suffering from conjunctivitis versus patients without ocular involvement, when treated with Dupilumab

ELIGIBILITY:
Inclusion Criteria:

* patients with severe atopic dermatitis resistant to main immunosuppressive drugs
* treated with Dupilumab
* with or without conjunctivitis
* postmenopausal women (since minimum 24 months), surgically sterilized women or women on contraception

Exclusion Criteria:

- pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Increase of lacrimal inflammatory cytokines | Month 8
  Change in inflammatory cytokines in tears collected by capillary before and after treatment with Dupilumab. Analysis will be performed by flow cytometry. Concentrations of the following cytokines wil be measured: interleukin-1 β, interleukin-3, interleukin-4, interleukin-5, interleukin-6, interleukin-8, interleukin-10, interleukin-13, interleukin-17, interferon α, Tumor Necrosis Factor α.

SECONDARY OUTCOMES:
Comparison of the increase of lacrimal inflammatory cytokines between the 2 groups | Month 8
  Change in inflammatory cytokines in tears collected by capillary among conjunctivitis patients versus non conjunctivitis patients, when treated with Dupilumab. Analysis will be performed by flow cytometry. Concentrations of the following cytokines wil be measured: interleukin-1 β, interleukin-3, interleukin-4, interleukin-5, interleukin-6, interleukin-8, interleukin-10, interleukin-13, interleukin-17, interferon α, Tumor Necrosis Factor α.
Absence/Presence of demodex | Day 0
  Presence of demodex on lashes before treatment with Dupilumab
Increase of lacrimal eosinophiles | Month 8
Improvement of quality of life | Month 8
  Improvement of quality of life for patients treated with Dupilumab, assessed with Ocular Surface Disease Index (OSDI) questionnaire, scored from 0 (normal/no ocular involvement) to 100 (severe ocular disease)

CONTACTS AND LOCATIONS:
Overall Officials: Camille FEBVAY, MD, Principal Investigator — CHU de Besançon

IPD SHARING:
Plan to Share IPD: No